CLINICAL TRIAL: NCT04589260
Title: A Ph 1, Rndmzd, Dbl-Blinded, Pbo-Controlled, 4-Part Study to Eval the Safety, Tolerability, PK, and PD of TD-1058 Admin by Inhalation of Single (A) and Multiple (B) Ascending Doses in Healthy Subjs and Subjs With IPF (C) and Following Admin Microtracer Doses (D)
Brief Title: TD-1058 First-In-Human Study in Healthy Subjects and Subjects With Idiopathic Pulmonary Fibrosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor has decided to stop the study due to business reasons. Study was terminated before initiation of part C and D (Decision to not proceed with Parts C and D was not for safety reasons and do not impact the overall risk benefit of the IMP.)
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0185; 2020-003003-34 (EudraCT Number)
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
Keywords: IPF; Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Fibrosis; Lung diseases, interstitial
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Fibrosis; Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blinded, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TD-1058 (Experimental): Part A (SAD): 6 out of 8 subjects per cohort (up to 5 cohorts) will be randomized to receive a single dose of TD-1058
  Part B (MAD): 6 out of 8 subjects per cohort (up to 4 cohorts) will be randomized to receive multiple dose of TD-1058
  Part C (IPF subjects): 8 out of 12 subjects per cohort (up to 2 cohorts) will be randomized to receive multiple dose of TD-1058
  Part D (Healthy Subjects): 6 subjects (1 cohort) will receive a single dose of TD-1058. After receipt of initial dose, subjects will recieve infusion of radiolabeled TD-1058 microtracer.
  Interventions: Drug: TD-1058
- Placebo (Placebo Comparator): Part A (SAD): 2 out of 8 subjects per cohort (up to 5 cohorts) will be randomized to receive a single dose of placebo
  Part B (MAD): 2 out of 8 subjects per cohort (up to 4 cohorts) will be randomized to receive multiple dose of placebo
  Part C (IPF subjects): 4 out of 12 subjects per cohort (up to 2 cohorts) will be randomized to receive multiple dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TD-1058 — Study drug to be administered by oral inhalation
  Arms: TD-1058
Drug: Placebo — Placebo to be administered by oral inhalation
  Arms: Placebo

SUMMARY:
This is a Phase 1, 4-part, randomized, double-blinded, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of TD-1058 inhaled solution. Part A is a SAD study in healthy subjects, Part B is a MAD study in healthy subjects, Part C is a multiple-dose study in subjects with IPF, and Part D studies lung bioavailability and renal elimination in Healthy Subjects.

DETAILED DESCRIPTION:
A Phase 1, 3-part, randomized, double-blinded, placebo-controlled, first in human study.

Part A is a single ascending dose (SAD) study in up to 5 cohorts of 8 healthy subjects (6 active and 2 placebo).

Part B is a multiple ascending dose (MAD) study in up to 4 cohorts of 8 healthy subjects (6 active and 2 placebo).

Part C is a 28 day multiple-dose study in up to 2 cohorts of 12 IPF subjects (8 active and 4 placebo). The dose levels administered in Part C will not exceed those previously administered in Part B which were shown to be well tolerated.

Part D studies lung bioavailability and renal elimination in Healthy Subjects.

ELIGIBILITY:
Inclusion Criteria:

Parts A and B:

* Healthy, adult, male or female, 18 to 60 years of age, inclusive, at Screening
* Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2 and weighs at least 50 kg at Screening
* Medically healthy with no clinically significant medical history, physical examination, spirometry, vital signs or ECGs, as deemed by the Investigator or designee
* Forced expiratory volume of 1 second (FEV1) ≥80% predicted at Screening and prior to dosing
* No clinically significant abnormalities in the results of laboratory evaluations at Screening and the visit scheduled between Day -7 and Day -2, as applicable, and at the discretion of the Investigator and Sponsor's Medical Monitor.
* Pregnancy concerns:

  * Female subjects must either of non-childbearing potential or if of childbearing potential, subject must not be pregnant or breastfeeding, and must agree to use a highly effective birth control method during the study and through 30 days after the last dose of study medication
  * Male subjects must agree to use condoms to prevent potential fetal or partner exposure through seminal fluid, in addition to the use of highly effective pregnancy prevention measures with female partners of childbearing potential during the study and through 30 days after the last dose of study medication
  * Subjects must agree to not donate ova or sperm through 30 days after the last dose of study medication
* Able to understand the correct technique for the use of the nebulizer device(s) at Screening, Day -1, and prior to dosing on Day 1, as applicable
* Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol
* Part B Only: Willing to undergo 2 bronchoscopy procedures and must be able to tolerate the bronchoscopy at Screening

Part C (Subjects with IPF):

* Male subjects ≥ 45 years and female subjects ≥ 55 years at Screening
* Body mass index (BMI) ≥ 18.0 and ≤ 35.0 kg/m2 and weighs at least 45 kg at Screening
* Diagnosis of IPF
* Forced expiratory vital capacity (FVC) > 50% predicted and diffusing capacity of the lungs for carbon monoxide (DLCO) > 35% predicted
* Subjects with IPF will be those who are not eligible for anti-fibrotic treatment according to NICE criteria or the subjects who are intolerant of or declined immediate commencement of standard first-line therapy with anti-fibrotics.
* Pregnancy concerns:

  * Female subjects must either of non-childbearing potential or if of childbearing potential, subject must not be pregnant or breastfeeding, and must agree to use a highly effective birth control method during the study and through 30 days after the last dose of study medication
  * Male subjects must agree to use condoms to prevent potential fetal or partner exposure through seminal fluid, in addition to the use of highly effective pregnancy prevention measures with female partners of childbearing potential during the study and through 30 days after the last dose of study medication
  * Subjects must agree to not donate ova or sperm through 30 days after the last dose of study medication
* Able to understand the correct technique for the use of the nebulizer device(s) at Screening, and prior to dosing on Day 1, as applicable

Part D (Microtracer):

* Healthy, adult, male, 18 to 60 years of age, inclusive, at Screening.
* BMI ≥ 18.0 and ≤ 30.0 kg/m2 at Screening and weighs at least 50 kg at Screening.
* Medically healthy with no clinically significant medical history, physical examination, spirometry, vital signs or ECGs, as deemed by the Investigator or designee.
* FEV1 ≥80% predicted at Screening and prior to dosing.
* No clinically significant abnormalities in the results of laboratory evaluations at Screening and Day -1, as applicable and at the discretion of the Investigator and Sponsor's Medical Monitor.
* Pregnancy concerns:

  * Male subjects must agree to use condoms to prevent potential fetal or partner exposure through seminal fluid, in addition to the use of highly effective pregnancy prevention measures with female partners of childbearing potential during the study and through 90 days after the last dose of study medication
  * Subjects must agree to not donate ova or sperm through 30 days after the last dose of study medication
* Able to understand the correct technique for the use of the nebulizer device(s) at Screening, and prior to dosing on Day 1, as applicable

Exclusion Criteria:

Parts A and B:

* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the Investigator or designee
* Abnormal ECG measurements at Screening (any of the three individual ECG measurements) or prior to dosing indicating a second- or third- degree atrioventricular block, or one or more of the following:

  * QRS > 120 msec
  * QTcF > 450 msec (males) or > 460 msec (females)
  * PR interval > 220 msec
* Known personal or family history of congenital long QT syndrome or known family history of sudden death.
* Supine resting bradycardia (pulse < 40 beats per minute [bpm]) or a supine resting tachycardia (pulse > 100 bpm) at Screening or prior to dosing on Day 1.
* Abnormal renal function as defined by estimated glomerular filtration rate (eGFR) <90mL/min/1.73m^2 at Screening
* History of clinically significant hypotensive episodes or symptoms of fainting, dizziness, or light-headedness.
* History or symptoms of clinically relevant neurologic disease, including transient ischemic attack, stroke, seizure disorder, or behavioral disturbances.
* History of lymphoma, leukemia, or other types of malignancy (except for completely resected squamous or basal cell cancer).
* Any signs of respiratory tract infection within 6 weeks of Screening that is deemed clinically significant by the Investigator and Sponsor's Medical Monitor.
* Has a current bacterial, parasitic, fungal, or viral infection; any infection requiring hospitalization or intravenous antibiotics within 6 months prior to Screening; any non respiratory tract infection requiring oral or topical antimicrobial treatment within 2 weeks prior to Screening; a history of more than one episode of herpes zoster infection.
* Subject has any condition of the oro-laryngeal or respiratory tract (including, but not limited to, prior surgery) that could possibly affect drug administration, deposition, or absorption, or ability to perform lung function measurements (spirometry), as determined by the Investigator or Sponsor.
* History or presence of alcoholism or drug abuse within the past 2 years prior to dosing.
* Positive urine drugs of abuse test result at Screening or Day -1.
* Positive urine or breath alcohol results at Screening or Day -1.
* Regular alcohol consumption of > 21 units per week for males or > 14 units per week for females, with one unit = ½ pint beer, a 25 mL shot of 40% spirit or a 125 mL glass of wine depending on type.
* Excessive caffeine intake (i.e., more than 5 cups of coffee/tea per day, or equivalent, on a regular basis).
* History of hypersensitivity to drugs, latex allergy, band aids, adhesive dressing, or medical tape, with a clinically significant reaction as determined by the Investigator or designee.
* History of severe allergic reaction (including anaphylaxis), or severe hypersensitivity or idiosyncratic reaction to any food, insect or bee sting, or previous status asthmaticus (e.g., acute severe asthma attacks).
* History or presence of hypersensitivity or idiosyncratic reaction to TD-1058, related compounds (e.g., ALK5 inhibitors), riboflavin or excipients, including severe milk protein allergy.
* Uses or has used tobacco or nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, patches etc.) within 6 months prior to Screening, or has a history of > 5 pack-years.
* Subject who has had a live viral vaccine (e.g., measles-mumps-rubella, varicella zoster, herpes zoster, oral polio virus, FluMist, attenuated typhoid fever vaccine, or attenuated rotavirus vaccine) within 8 weeks prior to Screening and/or is unwilling to avoid live viral vaccines for until at-least 8 weeks following completion of the final study visit.
* Positive results at Screening for human immunodeficiency virus (HIV), hepatitis A virus (HAV) antibodies (anti-HAV: both immunoglobulin (Ig)G and IgM positive, IgG positive in the absence of IgM positive is acceptable), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
* Subject who tests positive for active Coronavirus disease 2019 (COVID-19).
* Subject who has a history of latent or active tuberculosis, including positive QuantiFeron® Test result at Screening.
* Donation of blood (≥ 400 mL) or plasma, or significant blood loss within 56 days prior to the first dosing (including blood sampling requirement volumes from previous study participation)
* Participation in another clinical study (including medical device study) and received an investigational product within 90 days for small molecule drugs (or 5 half-lives of the investigational drug if longer than 90 days) or 60 days for biologics (or 5 half-lives of the investigational drug if longer than 60 days) prior to dosing. The 90 day / 60-day / 5 half lives window will be derived from the date of the last dosing in the previous study to Day 1 of the current study.
* Subject who, for any reason, is deemed by the Investigator to be inappropriate for this study; or has any condition which would confound or interfere with the evaluation of the safety, tolerability, or PK of the investigational drug; or is unable to comply with the study protocol.

Part C (Subjects with IPF):

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). ALT, AST, and total bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Abnormal ECG measurements at Screening (any of the three individual ECG measurements) or prior to dosing indicated by QTcF > 450 msec for males, QTcF > 460 msec for females.
* IPF exacerbation or upper or lower respiratory tract infection in the 8 weeks prior to dosing.
* Severe co-existent chronic obstructive pulmonary disease, for example FEV1 < 60% predicted.
* Currently taking Pirfenidone or Nintedanib or who have received Pirfenidone or Nintedanib within the 30 days prior to the first dosing on Day 1. Subjects using anti-fibrotic therapy as their standard of care treatment are not to be included in the study and must not withdraw existing IPF standard of care treatments in order to fulfil study eligibility criteria
* Prescribed long-term continuous home oxygen therapy (those whose use of oxygen is intermittent and for symptom relief only are not excluded).
* History of alcohol consumption regularly in excess of: An average weekly intake of > 21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (~125 ml) of wine or 1 (~25 ml) measure of spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 3 months prior to Screening.
* History of sensitivity to any of the study medications, or components thereof (i.e., riboflavin) or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation .
* Subject who has a history of latent or active tuberculosis , including positive QuantiFeron® Test result at Screening.
* Subject who tests positive for active COVID-19.
* A positive test for HIV antibody.
* Presence of HBsAg, positive hepatitis C antibody test result at Screening or within 3 months prior to first dose of study treatment. Subjects with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C ribonucleic acid (RNA) RT-PCR test is obtained.
* Positive urine drugs of abuse test result at Screening or Day 1.
* Positive urine or breath alcohol results at Screening or Day 1.
* Donation of blood (≥ 400 mL) or plasma, or significant blood loss within 56 days prior to the first dosing (including blood sampling requirement volumes from previous study participation).
* Participation in another clinical study (including medical device study) and received an investigational product within 90 days for small molecule drugs (or 5 half-lives of the investigational drug if longer than 90 days) or 60 days for biologics (or 5 half-lives of the investigational drug if longer than 60 days) prior to dosing. The 90-day / 60-day / 5 half-lives window will be derived from the date of the last dosing in the previous study to Day 1 of the current study.
* Participated in more than 4 clinical trials within 12 months prior to the first dosing on Day 1.
* Supine resting bradycardia (pulse < 40 beats per minute [bpm]) or a supine resting tachycardia (pulse > 100 bpm) at Screening
* Abnormal renal function as defined by eGRF < 60 mL/min/1.73m^2 at Screening
* History of lymphoma, leukemia, or other types of malignancy (except for completely resected squamous or basal cell cancer).
* Subject who has had a live viral vaccine (e.g., measles-mumps-rubella, varicella zoster, herpes zoster, oral polio virus, FluMist, attenuated typhoid fever vaccine, or attenuated rotavirus vaccine) within 8 weeks prior to Screening and/or is unwilling to avoid live viral vaccines for until at-least 8 weeks following completion of the final study visit.
* History or presence of hypersensitivity or idiosyncratic reaction to TD-1058, related compounds (e.g., ALK5 inhibitors), riboflavin or excipients, including severe milk protein allergy.
* Subject has previously received TD-1058.

Part D (Microtracer):

* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the Investigator or designee.
* Abnormal ECG measurements at Screening (any of the three individual ECG measurements) or prior to dosing indicating a second- or third- degree atrioventricular block, or one or more of the following:

  * QRS > 120 msec
  * QTcF > 450 msec
  * PR interval > 220 msec.
* Known personal or family history of congenital long QT syndrome or known family history of sudden death.
* Supine resting bradycardia (pulse < 40 bpm) or a supine resting tachycardia (pulse > 100 bpm) at Screening or prior to dosing on Day 1.
* History of clinically significant hypotensive episodes or symptoms of fainting, dizziness, or light-headedness.
* History or symptoms of clinically relevant neurologic disease, including transient ischemic attack, stroke, seizure disorder, or behavioral disturbances.
* History of lymphoma, leukemia, or other types of malignancy (except for completely resected squamous or basal cell cancer).
* Any signs of respiratory tract infection within 6 weeks of Screening that is deemed clinically significant by the Investigator and Sponsor's Medical Monitor.
* Has a current bacterial, parasitic, fungal, or viral infection; any infection requiring hospitalization or intravenous antibiotics within 6 months prior to Screening; any non-respiratory tract infection requiring oral or topical antimicrobial treatment within 2 weeks prior to Screening; a history of more than one episode of herpes zoster infection.
* Subject has any condition of the oro-laryngeal, naso-pharyngeal, or respiratory tract (including, but not limited to, prior surgery, e.g., nasal septal defects, perforation) that could possibly affect drug administration, deposition, or absorption, or ability to perform lung function measurements (spirometry), as determined by the Investigator or Sponsor.
* History or presence of alcoholism or drug abuse within the past 2 years prior to dosing.
* Positive urine drugs of abuse test result at Screening or Day -1.
* Positive urine or breath alcohol results at Screening or Day -1.
* Regular alcohol consumption of > 21 units per week, with one unit = ½ pint beer, a 25 mL shot of 40% spirit or a 125 mL glass of wine depending on type.
* Excessive caffeine intake (i.e., more than 5 cups of coffee/tea per day, or equivalent, on a regular basis).
* History of hypersensitivity to drugs, latex allergy, band aids, adhesive dressing, or medical tape, with a clinically significant reaction as determined by the Investigator or designee.
* History of severe allergic reaction (including anaphylaxis), or severe hypersensitivity or idiosyncratic reaction to any food, insect or bee sting, or previous status asthmaticus (e.g., acute severe asthma attacks).
* History or presence of hypersensitivity or idiosyncratic reaction to TD-1058, related compounds (e.g., ALK5 inhibitors), riboflavin or excipients, including severe milk protein allergy.
* Uses or has used tobacco or nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, patches etc.) within 6 months prior to Screening, or has a history of > 5 pack-years.
* Subject who has had a live viral vaccine (e.g., measles-mumps-rubella, varicella zoster, herpes zoster, oral polio virus, FluMist, attenuated typhoid fever vaccine, or attenuated rotavirus vaccine) within 8 weeks prior to Screening and/or is unwilling to avoid live viral vaccines for until at-least 8 weeks following completion of the final study visit.
* Positive results at Screening for HIV, HAV antibodies (anti-HAV: both IgG and IgM positive, IgG positive in the absence of IgM positive is acceptable), HBsAg or HCV.
* Subject who tests positive for active COVID-19.
* Subject who has a history of latent or active tuberculosis, including positive QuantiFeron® Test result at Screening.
* Subject is unable to refrain from or anticipates the use of any medication, herbal remedies, or vitamin supplements
* Subject has dietary restrictions incompatible with the diet that can be provided by the study site, in the opinion of the Investigator or designee or is unwilling to refrain from consuming restricted foods and beverages during the study
* Donation of blood (≥ 400 mL) or plasma, or significant blood loss within 56 days prior to the first dosing (including blood sampling requirement volumes from previous study participation.
* Donation of bone marrow within the last 6 months prior to dosing.
* Participation in another clinical study (including medical device study) and received an investigational product within 90 days. The 90-day window will be derived from the date of the last dosing in the previous study to Day 1 of the current study.
* Subject for whom the radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeds 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation (Medical Exposure) Regulations 2017 [23], shall participate in the study.
* Subjects who have been administered an investigational medicinal product in an absorption, metabolism, and excretion study in the last 12 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Part A (SAD) - Adverse Events | Part A (SAD) Day 1 to Day 8
  Number and severity of treatment emergent adverse events
Part B (MAD) - Adverse Events | Part B (MAD) Day 1 to Day 21
  Number and severity of treatment emergent adverse events
Part C (IPF) - Adverse Events | Part C (IPF) Day 1 to Day 35
  Number and severity of treatment emergent adverse events
Part D (Microtracer) - Adverse Events | Part D (Microtracer) Day 1 to Day 8
  Number and severity of treatment emergent adverse events

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of TD-1058: AUC | Part A (SAD) Day 1 to Day 8 Part B (MAD) Day 1 to Day 21 Part C (IPF) Day 1 to Day 35 Part D (Microtracer) Day 1 to Day 8
  Multiple PK variables of TD-1058 will be assessed during Part A, B, C and D and may include, but are not limited to: Area under the plasma concentration-time curve (AUC)
Pharmacokinetics (PK) of TD-1058: Cmax | Part A (SAD) Day 1 to Day 8 Part B (MAD) Day 1 to Day 21 Part C (IPF) Day 1 to Day 35 Part D (Microtracer) Day 1 to Day 8
  Multiple PK variables of TD-1058 will be assessed during Part A, B and C and may include, but are not limited to: Maximum observed concentration (Cmax)
Pharmacokinetics (PK) of TD-1058: Tmax | Part A (SAD) Day 1 to Day 8 Part B (MAD) Day 1 to Day 21 Part C (IPF) Day 1 to Day 35 Part D (Microtracer) Day 1 to Day 8
  Multiple PK variables of TD-1058 will be assessed during Part A, B and C and may include, but are not limited to: Time to reach maximum observed concentration (Tmax)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Theravance Biopharma Investigational Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.